CLINICAL TRIAL: NCT01514396
Title: Evaluation of Surgiseal as a Topical Emergency Department Skin Incision Adhesive in Pediatrics A Case Series
Brief Title: Skin Incision Adhesive in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R11-018
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2017-08

CONDITIONS: Wounds
Keywords: Pediatric; Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical Glue (Experimental): Surgiseal
  Interventions: Device: Surgiseal

INTERVENTIONS:
Device: Surgiseal — surgical glue

SUMMARY:
The purpose of this study is to evaluate the effectiveness of on-label use of Surgiseal™ Tissue Adhesive, a cyanoacrylate-based Surgical Topical Skin Tissue Adhesive in wound closure of the topical skin in children presenting in the Emergency Department (ED).

DETAILED DESCRIPTION:
Subjects had SurgiSeal™ applied to their topical skin incisions in the ED. Subjects' wounds were evaluated for bleeding and closure of the incision/wound before patient discharge and 48 hours after the procedure. Further follow up wound closure evaluations were conducted via telephone interview at 5-10 days and 14 days after the ED visit.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 5 and 18 years of age, inclusive
* Candidate for use of a topical surgical skin adhesive
* Informed consent by a parental guardian

Exclusion Criteria:

* A wound with evidence of active infection or gangrene or wounds of decubitus etiology
* Mucosal surfaces or across mucocutaneous junctions or skin that might be exposed to body fluids or dense natural hair
* Subjects with known hypersensitivity to cyanoacrylate or formaldehyde

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Drower, MS, Study Director — Medline Industries
Locations (1):
- Akron Children's Hospital Emergency Department, Akron, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgical Glue: Surgiseal
  Surgiseal: surgical glue To determine if SurgiSeal™ can effectively seal epidermal wounds in children while not causing any adverse events.
Period: Overall Study
Arm/Group | Surgical Glue
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Surgical Glue
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Closure
Description: wound closure measured baseline to 14 days
Time Frame: baseline to 14 days
Measure: Number; unit: participants
Groups:
- Wound Closure: Number of Participants with Wound Closure baseline to 14 days from discharge
Arm/Group | Wound Closure
Number analyzed (Participants) | 8
participants | 8

2. Secondary Outcome: Adverse Events Related to Wound Closure
Description: Adverse events reported
Time Frame: 14 days
Measure: Number; unit: participants
Groups:
- Adverse Events Related to Wound Closure: Adverse Events related to wound closure with study product
Arm/Group | Adverse Events Related to Wound Closure
Number analyzed (Participants) | 8
participants | 0

ADVERSE EVENTS:
Time Frame: baseline to 14 days
Arm/Group | Surgical Glue
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No